CLINICAL TRIAL: NCT04020913
Title: Recombinant Human Growth Hormone (GH): Effects on Metabolic Profile, Body Composition and Skeletal Muscle Strength and Function in Pre-pubertal Short Boys With and Without GH Deficiency
Brief Title: Skeletal Muscle Effects of GH in Boys
Status: Completed | Type: Observational
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Nelly Mauras, MD, Nemours Children's Clinic
Other Study IDs: #19-09; U111112218502 (Other Grant/Funding Number: Novo Nordisk)
Record Dates: First submitted 2019-05-24; First posted 2019-07-16 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Growth Hormone Deficiency; Idiopathic Short Stature
Keywords: GH; muscle strength; prepubertal; boys; short stature; GH treatment; muscle agility
MeSH Terms: conditions — Dwarfism, Pituitary; Dwarfism | interventions — Human Growth Hormone; Growth Hormone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum/plasma will be obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Short Stature Boys: Prepubertal boys with short stature defined as a height ≤-2 SDS with either GH deficiency (defined as peak GH responses to pharmacologic stimuli <10ng/ml) or idiopathic short stature (i.e., no identifiable pathology) will be studied pre and post 12 months of GH therapy.
  Interventions: Drug: Somatropin injection
- Normally Statured Boys: A group of 15 healthy, normally statured (between 10th- 90th %), age-matched boys not on Growth Hormone replacement, preferably siblings (although not exclusively), will be recruited to serve as healthy controls.

INTERVENTIONS:
Drug: Somatropin injection — Boys with short stature will be studied for measures of:
  1. skeletal muscle strength, power, and endurance
  2. muscle agility
  3. lean body mass accrual
  4. bone mineral density and resting energy expenditure before and after 6 months and 12 months of GH administration
  Other Names: Recombinant Growth Hormone; Norditropin
  Groups: Short Stature Boys

SUMMARY:
The purpose of the study is to measure the functional effects of recombinant GH in skeletal muscle, in addition to growth promotion, in short prepubertal boys with either growth hormone deficiency or idiopathic short stature. Patients will be similarly short. The investigators will also compare these values in the short stature cohort to those obtained in testing performed in normally growing age-matched healthy control boys not on GH. The group on GH will be studied before and after 6 and 12 months of GH treatment.

DETAILED DESCRIPTION:
Prepubertal boys with significant short stature (height SDS ≤-2.0) diagnosed with either GH deficiency or idiopathic short stature (ISS) who are identified as candidates for GH treatment will recruited. Subjects will have a battery of studies to assess skeletal muscle strength, agility, power and endurance, as well as assessment of body composition and energy expenditure before and after GH administration. GH (Somatropin) treatment at standard doses will be given as daily injections at bedtime. Subjects will be followed at three-month intervals per the clinical routine, when anthropometric measurements will be obtained. Baseline studies will be repeated at 6 and 12 months from initiation of treatment, each patient will serve as his own control pre and post GH.

A group of normally statured healthy boys will have the same testing as the study patients but without GH treatment to assess the impact of natural growth on the muscle measures above.

ELIGIBILITY:
Inclusion Criteria:

Short Stature Group

1. 30 boys between 6-11 years of age
2. Prepubertal
3. Short stature (height ≤ -2SDS) due to either GH deficiency or idiopathic
4. Stable treatment of other pituitary hormone deficiencies
5. Naïve to GH therapy, or GH discontinued at least 6 months prior to study

Normal Stature Group

1. 15 boys between 6-11 years of age
2. Prepubertal
3. Normal height (10th to 90th%)

Exclusion Criteria:

1. Actively growing brain tumors
2. Chronic medical conditions that could affect study outcomes
3. Long-term steroid use
4. Intense regular physical training programs or organized team sports

Ages: 6 Years to 11 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Prepubertal boys with short stature defined as a height ≤-2 SDS with either GH deficiency (i.e., peak GH responses to pharmacologic stimuli <10ng/ml) or idiopathic short stature (i.e., normal GH, no identifiable pathology) will be studied.
  Normally Statured Boys: A group of 15 healthy, normally statured (between 10th- 90th %), age-matched boys not on somatropin, preferably siblings (although not exclusively) will be studied similarly.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle strength (Newtons) | 12 months
  Upper and lower body muscle strength will be assessed using a handheld dynamometer for manual muscle testing of peak force

SECONDARY OUTCOMES:
Skeletal muscle power (Watts) | 12 months
  Lower extremity power will be assessed by vertical jump performed using a Power time mat
Muscle agility (seconds) | 12 months
  Muscle agility will be assessed by a timed shuttle run
Muscle endurance | 12 months
  Upper body muscular endurance will be assessed using a modified push up test for repetitions
Lean body mass accrual | 12 months
  Assessed by dual energy x-ray absorptiometry (DEXA) scan of the whole body
Bone mineral density | 12 months
  Assessed by DEXA scan of the lumbar spine and whole body
Resting energy expenditure | 12 months
  Indirect calorimetry will be performed after overnight fast

CONTACTS AND LOCATIONS:
Overall Officials: Nelly Mauras, MD, Principal Investigator — Nemours Children's Clinic
Locations (1):
- Nemours Children's Clinic, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No